CLINICAL TRIAL: NCT03123120
Title: Proof-of-concept Study of BI 655130 add-on Treatment in Patients With Mild-to-moderately Active Ulcerative Colitis During TNF Inhibitor Therapy
Brief Title: A Study in Patients With Mild or Moderate Ulcerative Colitis Who Take a TNF Inhibitor. The Study Investigates Whether Bowel Inflammation Improves When Patients Take BI 655130 in Addition to Their Current Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1368-0010; 2016-004572-21 (EudraCT Number)
Record Dates: First submitted 2017-04-13; First posted 2017-04-21 (Actual); Results first posted 2021-10-07 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — spesolimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spesolimab (Experimental): 1200 milligrams (mg) of Spesolimab (BI 655130) were administered every 4 weeks (q4w) via intravenous infusion over 12 weeks of treatment (3 injections of Spesolimab 1200 mg in total during the 12 weeks: at Week 0, 4, and 8 respectively).
  Interventions: Drug: Spesolimab
- Placebo (Placebo Comparator): Matching placebo was administered via intravenous infusion over 12 weeks of treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spesolimab — 12 weeks treatment
  Other Names: BI 655130
  Arms: Spesolimab
Drug: Placebo — 12 weeks treatment
  Arms: Placebo

SUMMARY:
The objectives of this trial are safety and efficacy (proof-of-concept) of induction of mucosal healing by BI 655130 add-on therapy in patients with mild or moderate ulcerative colitis and persisting endoscopic activity despite pre-existing TNFi treatment.

This trial will explore safety and efficacy of a dose of BI 655130 that was modelled to achieve the similar exposures as the highest exposures tested and found safe and tolerable in preceding single and multiple dose studies in healthy subjects, as add-on to pre-existing TNFi (Tumor necrosis factor inhibitor) treatment. Secondary and further objectives include assessment of the pharmacokinetic (PK) profile of BI 655130 and early exploration of specific biomarkers with potential usefulness to predict clinical efficacy or safety outcome or help understand BI 655130's mode of action.

ELIGIBILITY:
Inclusion Criteria

* 18 - 75 years at screening and randomisation
* Diagnosis of ulcerative colitis >= 5 months prior to screening
* Receiving TNFi treatment with doses (i.e. dose and dosing interval) unchanged for >= 4 months (Infliximab) or >= 2 Monaten (Adalimumab or Golimumab) prior to randomisation
* Mild or moderate disease activity, defined as total Mayo Score (MCS) (<= 10)
* Further inclusion criteria apply

Exclusion Criteria:

* Prior use of more than two different TNF inhibitors or vedolizumab
* Extensive colonic resection
* Evidence of infection with C. difficile or other intestinal pathogen <28 days prior to screening
* Active or latent tuberculosis
* Further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-09-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- Denmark (3):
  - Aalborg Sygehus Syd, Aalborg
  - Sanos Clinic, Herlev
  - Odense University Hospital, Odense
- Germany (5):
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Ulm, Ulm
- Amsterdam UMC, Locatie AMC, Amsterdam, Netherlands
- Akershus Universitetssykehus HF, Lørenskog, Norway
- Spain (3):
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Politècnic La Fe, Valencia
- United Kingdom (3):
  - St James's University Hospital, Leeds
  - Guy's Hospital, London
  - Whiston Hospital, Prescot

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Lebwohl MG, Thoma C, Haeufel T. Spesolimab use in generalised pustular psoriasis flares - Authors' reply. Lancet. 2024 Aug 31;404(10455):847-848. doi: 10.1016/S0140-6736(24)01557-5. No abstract available. PMID 39216969
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized, placebo-controlled, double-blind, parallel-group trial over 36 weeks, including a 24-week follow-up period evaluated safety and efficacy of induction of mucosal healing by Spesolimab (BI 655130) add-on therapy in patients with mild or moderate ulcerative colitis and persisting endoscopic activity despite pre-existing tumor necrosis factor inhibitor treatment.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo - Randomized: Matching placebo was administered via intravenous infusion over 12 weeks of treatment.
  Participants who were randomized into the Placebo treatment were included in this arm.
- Spesolimab 1200 mg - Randomized: 1200 milligrams (mg) of Spesolimab (BI 655130) were administered every 4 weeks (q4w) via intravenous infusion over 12 weeks of treatment (3 injections of Spesolimab 1200 mg in total during the 12 weeks: at Week 0, 4, and 8 respectively).
  Participants who were randomized into the Spesolimab 1200 mg treatment were included in this arm.
Period: Overall Study
Arm/Group | Placebo - Randomized | Spesolimab 1200 mg - Randomized
Started | 8 | 14
Safety Analysis Set (SAF) (1 patient who was randomized to placebo accidentally received one dose of Spesolimab and was analyzed in the Spesolimab group in the SAF) | 7 | 15
Completed (Completed planned observation time.) | 8 | 12
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): This patient set includes all patients in the safety analysis set who had a baseline measurement available for the primary endpoint. Treatment assignment will be as randomized. Patients who were randomized but not treated were excluded from the FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - Randomized | Spesolimab 1200 mg - Randomized | Total
Number analyzed (Participants) | 8 | 14 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.5 (12.1) | 43.1 (9.9) | 44.0 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 7 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 14 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 13 | 21
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Mayo clinical score (MCS) modified endoscopic subscore (mESS) [Mean (Standard Deviation); unit: Score on a scale] — The Mayo clinical score (MCS) modified endoscopic subscore (mESS) at baseline was reported. The MCS mESS ranged from 0 (normal) to 3 (severe disease). The MCS mESS was assessed by a central reader who was independent from the investigator.
  Score on a scale | 2.8 (0.5) | 2.8 (0.4) | 2.8 (0.4)
Number of participants per Mayo clinical score modified endoscopic subscore value group [Count of Participants; unit: Participants] — The number of participants per Mayo clinical score (MCS) modified endoscopic subscore (mESS) value group was reported. The MCS mESS ranged from 0 (normal) to 3 (severe disease). The MCS mESS was assessed by a central reader who was independent from the investigator.
  Participants
    0 | 0 | 0 | 0
    1 | 0 | 0 | 0
    2 | 2 | 3 | 5
    3 | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Endoscopic Improvement (MCS mESS ≤1) at Week 12
Description: Proportion of participants with endoscopic improvement (Mayo clinical score (MCS) modified endoscopic sub-score (mESS) ≤1) at Week 12 was reported. The endoscopic improvement (mucosal healing) was defined as the Mayo clinical score (MCS) modified endoscopic sub-score (mESS) ≤ 1 point. The MCS mESS ranged from 0 (normal) to 3 (severe disease). The mESS was assessed by a central reader who was independent from the investigator. The 95% confidence intervals (in the descriptive statistics part) were calculated using the method of Wilson.
Time Frame: At Week 12
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo - Randomized | Spesolimab 1200 mg - Randomized
Number analyzed (Participants) | 8 | 14
Proportion of participants | 0.375 [0.137 to 0.694] | 0.143 [0.040 to 0.399]
Statistical Analysis 1: Comparison: Placebo - Randomized vs Spesolimab 1200 mg - Randomized; Test type: Other; Risk Difference (RD) = -0.232, 95% CI 2-sided [-0.568 to 0.118] — Risk difference was calculated as the observed proportion of response from Spesolimab minus the one from Placebo. Newcombe method was used in the calculation of the 95% confidence interval around the risk difference

2. Secondary Outcome: Proportion of Participants With Total Clinical Remission (tCR) Based on Total Mayo Clinical Score at Week 12
Description: Proportion of participants with total clinical remission based on total Mayo clinical score at Week 12 was reported. The total clinical remission based on total Mayo clinical score was defined as the total Mayo clinical score ≤ 2 points and all sub-scores ≤ 1 point.
  The total Mayo clinical score was a composite disease activity score consisting of 4 sub-scores: stool frequency, rectal bleeding, physician's global assessment, and modified endoscopic appearance. Each sub-score ranged from 0 (normal) to 3 (severe disease/worse disease status). The total Mayo score was by summing up the four sub-scores and ranged from 0 to 12 with higher score indicating worse disease.
  The 95% confidence intervals (in the descriptive statistics part) were calculated using the method of Wilson.
Time Frame: At Week 12
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo - Randomized | Spesolimab 1200 mg - Randomized
Number analyzed (Participants) | 8 | 14
Proportion of participants | 0.125 [0.022 to 0.471] | 0.071 [0.013 to 0.315]
Statistical Analysis 1: Comparison: Placebo - Randomized vs Spesolimab 1200 mg - Randomized; Test type: Other; Risk Difference (RD) = -0.054, 95% CI 2-sided [-0.404 to 0.210] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Proportion of Participants With Histological Remission at Week 12
Description: Proportion of participants with histological remission at Week 12 was reported. The histological remission was defined as the Robarts histology index score ≤ 6.
  The Robarts histopathology index (RHI) was a histologic activity score, scoring the components chronic inflammatory infiltrate, lamina propria neutrophils, neutrophils in epithelium and erosion or ulceration on a scale of 0 to 3. The 4 components were weighted differently to calculate the RHI, with RHI = 1 × chronic inflammatory infiltrate level + 2 × lamina propria neutrophils + 3 × neutrophils in epithelium + 5 × erosion or ulceration. The resulting RHI score ranged from 0 (no disease activity) to 33 (severe disease activity).
  The 95% confidence intervals (in descriptive statistics part) were calculated using the method of Wilson.
Time Frame: At Week 12
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo - Randomized | Spesolimab 1200 mg - Randomized
Number analyzed (Participants) | 8 | 14
Proportion of participants | 0.500 [0.215 to 0.785] | 0.214 [0.076 to 0.476]
Statistical Analysis 1: Comparison: Placebo - Randomized vs Spesolimab 1200 mg - Randomized; Test type: Other; Risk Difference (RD) = -0.286, 95% CI 2-sided [-0.602 to 0.101] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Proportion of Participants With Clinical Remission (CR) Based on Mayo Clinical Score at Week 12
Description: Proportion of participants with clinical remission (CR) based on Mayo clinical score at Week 12 was reported. The clinical remission based on Mayo clinical score was defined as the total Mayo clinical Score ≤ 2 and Rectal Bleeding Subscore = 0, Stool Frequency Score =0 or 1 and drop ≥ 1 from baseline, and Modified endoscopic sub-score (mESS) ≤ 1.
  The total Mayo clinical score was a composite disease activity score consisting of 4 sub-scores: stool frequency, rectal bleeding, physician's global assessment, and modified endoscopic appearance. Each sub-score ranged from 0 (normal) to 3 (severe disease/worse disease status). The total Mayo clinical score was by summing up the four sub-scores and ranged from 0 to 12 with higher score indicating worse disease.
  The 95% confidence intervals (in the descriptive statistics part) were calculated using the method of Wilson.
Time Frame: At Week 12
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo - Randomized | Spesolimab 1200 mg - Randomized
Number analyzed (Participants) | 8 | 14
Proportion of participants | 0.000 [0.000 to 0.324] | 0.143 [0.040 to 0.399]
Statistical Analysis 1: Comparison: Placebo - Randomized vs Spesolimab 1200 mg - Randomized; Test type: Other; Risk Difference (RD) = 0.143, 95% CI 2-sided [-0.197 to 0.399] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with any treatment-emergent adverse events (TEAEs) was reported.
Time Frame: From first does of study medication until end of the follow-up period, up to 36 weeks.
Population: Safety Analysis Set (SAF): this patient set included all randomized patients who received at least one dose of trial drug. Treatment assignment was analyzed according to the actual treatment. 1 patient who was assigned to placebo accidentally received one dose of Spesolimab and was analyzed in the Spesolimab group in the SAF.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo - Actual: Matching placebo were administered via intravenous over 12 weeks of treatment. Participants who actually administered placebo during the study were included in this group. 1 patient who was assigned to placebo accidentally received one dose of Spesolimab and was analyzed in the Spesolimab group.
- Spesolimab 1200 mg - Actual: 1200 milligrams (mg) of Spesolimab (BI 655130) were administered every 4 weeks (q4w) via intravenous infusion over 12 weeks of treatment.
  Participants who actually administered Spesolimab during the study were included in this group. 1 patient who was assigned to Placebo accidentally received one dose of Spesolimab and was analyzed in the Spesolimab group.
Arm/Group | Placebo - Actual | Spesolimab 1200 mg - Actual
Number analyzed (Participants) | 7 | 15
Participants | 6 | 15

ADVERSE EVENTS:
Time Frame: From first does of study medication until end of the follow-up period, up to 36 weeks.
Description: Safety Analysis Set (SAF): this patient set included all randomized patients who received at least one dose of trial drug. Treatment assignment was analyzed according to the actual treatment. 1 patient who was assigned to placebo accidentally received one dose of Spesolimab and was analyzed in the Spesolimab group in the SAF.
Arm/Group | Placebo - Actual | Spesolimab 1200 mg - Actual
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/7 | 2/15
Other Adverse Events (participants affected / at risk) | 6/7 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Actual (N=7) | Spesolimab 1200 mg - Actual (N=15)
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Actual (N=7) | Spesolimab 1200 mg - Actual (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Episcleritis (Eye disorders) | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Influenza like illness (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Helicobacter gastritis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 4
Migraine (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT03123120/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT03123120/SAP_001.pdf